CLINICAL TRIAL: NCT01364649
Title: A Randomized, Double-Blind, Parallel-Group, Active-Controlled, Flexible-Dose Study Evaluating the Effect of Lu AA21004 vs Escitalopram on Sexual Functioning in Adults With Well-Treated Major Depressive Disorder Experiencing Selective Serotonin Reuptake Inhibitor-Induced Sexual Dysfunction
Brief Title: Vortioxetine (Lu AA21004) 10 and 20 mg for Treatment of Major Depressive Disorder With Sexual Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004_318; U1111-1120-3483 (Registry Identifier: WHO)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Treatment Outcome
Keywords: Sexual Dysfunction, Physiological; Depressive Disorder, Major; Depression; Antidepressive Agents; Drug Therapy
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Depressive Disorder, Major; Depression | interventions — Vortioxetine; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vortioxetine (Experimental): Vortioxetine 10 mg, tablets, orally, once daily for 1 week, then dose adjustment to a maximum 20 mg, tablets, orally, once daily for up to 7 weeks. At week 8, vortioxetine placebo-matching capsules, orally, once daily for 1 week only.
  Interventions: Drug: Vortioxetine; Drug: Placebo
- Escitalopram (Active Comparator): Escitalopram 10 mg, tablets, orally, once daily for 1 week, then escitalopram dose adjustment to a maximum 20 mg, capsules, orally, once daily for up to 7 weeks. At week 8, escitalopram 10 mg, capsules, capsules, orally, once daily for 1 week only.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine tablets
  Other Names: Lu AA21004
  Arms: Vortioxetine
Drug: Escitalopram — Escitalopram tablets
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — Vortioxetine Placebo-matching capsules
  Arms: Vortioxetine

SUMMARY:
The purpose of this study is to evaluate the effects of Vortioxetine (Lu AA21004), once daily (QD), compared with escitalopram on sexual functioning.

DETAILED DESCRIPTION:
The drug being tested in this study is called Lu AA21004. Lu AA21004 is being tested to treat people who have major depressive disorder (MDD). This study will look at sexual function in people who take Lu AA21004.

The study will enroll approximately 440 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Lu AA21004 10 to 20 mg
* Escitalopram 10 to 20 mg - This is a comparator drug that is also used to treat MDD.

All participants will be asked to take one tablet at the same time each day throughout the study. All participants will be asked to answer questionnaires at each study visit.

This multi-centre trial will be conducted in the United States and Canada. The overall time to participate in this study is 14 weeks. Participants will make 7 visits to the clinic, and will be contacted by telephone 21 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a man or a woman aged between 18 and 55 years, inclusive, who is currently being treated with selective serotonin reuptake inhibitor (SSRI) monotherapy (only citalopram, paroxetine, or sertraline allowed) for at least 8 weeks, which was prescribed to treat a major depressive episode (MDE), according to the DSM-IV-TR criteria.
2. Is currently stable; and has a Clinical Global Impression Scale-Severity of Illness Scale (CGI-S) score of ≤3.
3. Is currently experiencing treatment-emergent sexual dysfunction (TESD; defined as a Changes in Sexual Functioning Questionnaire (CSFQ-14) total score ≤41 for women and ≤47 for men), considered to be attributable to the current SSRI monotherapy and is suitable for a switch.

Exclusion Criteria:

1. Has previously participated in a Lu AA21004 clinical study.
2. Has 1 or more the following: any current psychiatric disorder other than MDD as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR; as assessed by the Mini International Neuropsychiatric Interview Version 6.0.0); current or history of manic or hypomanic episode, schizophrenia, or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR; current diagnosis of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in sustained full remission for at least 2 years prior to Screening (subject must also have negative urine drug screen prior to Baseline); presence or history of a clinically significant neurological disorder (including epilepsy); neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc); or any Axis II disorder that might compromise the study.
3. Has sexual dysfunction associated with an etiology other than SSRI treatment or current MDE (e.g., due to a medical condition, such as diabetes or hypertension, a medication, a genital anatomical deformity, or alcohol abuse).
4. Is nonsexually active or anticipates decreasing frequency of sexual activity (ie, sexual activity anticipated to lead to orgasm or that would normally lead to orgasm, which can include sexual intercourse, oral sex, masturbation, sexual fantasies, and/or thinking of sexual activity) during the course of the study below the level at study initiation.
5. Is a male with a history of premature ejaculation in the past year.
6. Has had major relationship changes during the preceding SSRI treatment period or plans to have major relationship changes during the course of the study.
7. Has a sexual partner(s) who plans to initiate treatment for sexual dysfunction during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 447 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Takeda
Locations (62):
- United States (53):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Anaheim, California
  - Chino, California
  - Costa Mesa, California
  - Encino, California
  - Escondido, California
  - Irvine, California
  - Newport Beach, California
  - Oceanside, California
  - San Diego, California
  - Norwich, Connecticut
  - Washington D.C., District of Columbia
  - Coral Springs, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Lauderhill, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Sanford, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Joliet, Illinois
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Gaithersburg, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Weymouth, Massachusetts
  - Flowood, Mississippi
  - Creve Coeur, Missouri
  - St Louis, Missouri
  - Toms River, New Jersey
  - Willingboro, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Charlottesville, Virginia
  - Seattle, Washington
  - Waukesha, Wisconsin
- Canada (9):
  - Medicine Hat, Alberta
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - Sydney, Nova Scotia
  - Burlington, Ontario
  - Chatham, Ontario
  - Kingston, Ontario
  - Mississauga, Ontario
  - Toronto, Ontario

REFERENCES:
- [Derived] Jacobsen PL, Nomikos GG, Zhong W, Cutler AJ, Affinito J, Clayton A. Clinical implications of directly switching antidepressants in well-treated depressed patients with treatment-emergent sexual dysfunction: a comparison between vortioxetine and escitalopram. CNS Spectr. 2020 Feb;25(1):50-63. doi: 10.1017/S1092852919000750. PMID 31010445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 57 sites in the US and 9 sites in Canada from 16 June 12011 to 9 December 2013.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 2 (flexible doses of either vortioxetine (Lu AA21004) 10/20 mg once daily (QD) or escitalopram 10/20 mg QD) treatment groups.
Groups:
- Vortioxetine: Vortioxetine 10 mg, tablets, orally, once daily for 1 week, then dose adjustment to a maximum 20 mg tablets, orally, once daily for up to 7 weeks. At week 8, vortioxetine placebo-matching capsules, orally, once daily for 1 week only.
Period: Overall Study
Arm/Group | Vortioxetine | Escitalopram
Started | 225 | 222
Completed | 169 | 179
Not Completed | 56 | 43
Not completed — Pretreatment Event or Adverse Event | 20 | 14
Not completed — Lack of Efficacy | 6 | 0
Not completed — Non-compliance with Investigational Drug | 1 | 0
Not completed — Protocol Deviations | 4 | 8
Not completed — Withdrawal of Consent | 9 | 7
Not completed — Lost to Follow-up | 12 | 13
Not completed — Other | 4 | 1

BASELINE CHARACTERISTICS:
Population: All randomized set (N=447): All study participants who were screened and randomized to one of two treatment arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine | Escitalopram | Total
Number analyzed (Participants) | 225 | 222 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (9.96) | 40.2 (10.01) | 39.8 (9.98)
Age, Customized [Number; unit: participants]
  ≤41 years | 122 | 112 | 234
  >41 years | 103 | 110 | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 135 | 263
  Male | 97 | 87 | 184
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14 | 36 | 50
  Non-Hispanic and Non-Latino | 211 | 186 | 397
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (or White, including Hispanic) | 178 | 181 | 359
  Black of African American | 41 | 35 | 76
  Asian | 4 | 3 | 7
  American Indian or Alaska Native | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  North America | 225 | 222 | 447
Height [Mean (Standard Deviation); unit: cm] | 169.6 (9.73) | 170.3 (8.81) | 169.9 (9.28)
Weight [Mean (Standard Deviation); unit: kg] | 79.62 (16.202) | 81.22 (16.012) | 80.41 (16.110)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.54 (4.352) | 27.90 (4.440) | 27.72 (4.395)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 90.85 (13.274) | 93.31 (13.074) | 92.07 (13.218)
Smoking Classification [Number; unit: participants]
  Never smoked | 112 | 126 | 238
  Current smoker | 69 | 55 | 124
  Ex-smoker | 44 | 41 | 85
Alcohol Consumption [Number; unit: participants]
  Never | 65 | 65 | 130
  Once monthly or less often | 86 | 82 | 168
  Once a week | 40 | 37 | 77
  2 to 6 times per week | 33 | 36 | 69
  Daily | 1 | 2 | 3
Changes in Sexual Functioning Questionnaire Short-Form (CSFQ-14) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The CSFQ-14 is a structured self reported questionnaire designed to measure illness- and medication-related changes in sexual functioning consisting of 14 items that measure sexual functioning as a total score (14 items) and on the subscales of pleasure (1 item), desire/frequency (2 items), desire/interest (3 items), arousal (3 items), and orgasm (3 items), rated on an 5 point scale from 1 to 5 with a total score range from 14 to 70. Higher scores reflect higher sexual functioning. The number of participants with available data were 220 and 216 in each treatment arm respectively.
  scores on a scale | 36.5 (5.81) | 36.3 (5.62) | 36.4 (5.71)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). The number of participants with available data were 224 and 221 in each treatment arm respectively.
  scores on a scale | 7.9 (6.28) | 8.3 (6.53) | 8.1 (6.40)
Clinical Global Impression - Severity scale (CGI-S) score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. The number of participants with available data were 224 and 221 in each treatment arm respectively.
  scores on a scale | 2.0 (0.81) | 2.0 (0.84) | 2.0 (0.82)
Profile of Mood States (POMS) Brief Total Score [Mean (Standard Deviation); unit: scores on a scale] — POMS brief is a rating scale, which comprises of 30 items that are evaluated in a 0-4 scale (0=not at all and 4=extremely). The scores for the 30 items are added in various combinations to throw six validated factors which are used to calculate total POMS score: (tension-anxiety) + (depression-dejection) + (anger-hostility)+ (fatigue-Inertia) + (confusion-bewilderment) - (vigor-activity). Score range (-40 to 192). Score -40 denotes the best score and score 192 denotes the worst score. The number of participants with available data were 224 and 219 in each treatment arm respectively.
  scores on a scale | 18.8 (19.36) | 19.7 (19.45) | 19.2 (19.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Changes in Sexual Functioning Questionnaire Short-Form (CSFQ-14) Total Score at Week 8
Description: The CSFQ-14 is a structured self reported questionnaire designed to measure illness- and medication-related changes in sexual functioning consisting of 14 items that measure sexual functioning as a total score (14 items) and on the subscales of pleasure (1 item), desire/frequency (2 items), desire/interest (3 items), arousal (3 items), and orgasm (3 items), rated on an 5 point scale from 1 to 5 with a total score range from 14 to 70. Higher scores reflect higher sexual functioning. A positive change from Baseline indicates that symptoms have improved. The primary analysis was based on a mixed model for repeated measurements (MMRM) analysis of covariance with treatment, center, week, treatment-by-week interaction as fixed effects, Baseline CSFQ-14 total score-by-week as covariate, and a completely unstructured covariance matrix.
Time Frame: Baseline, Week 8
Population: Participants from the Full Analysis Set (FAS), defined as all participants who were randomized and received at least 1 dose of study drug, who had data available for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vortioxetine | Escitalopram
Number analyzed (Participants) | 165 | 173
scores on a scale | 8.8 (0.64) | 6.6 (0.64)
Statistical Analysis 1: Comparison: Vortioxetine vs Escitalopram; Test type: Superiority or Other; p = 0.013, Mixed Model Repeated Measurements; The primary analysis was performed by using observed case data only; LS mean difference = 2.2, 95% CI 2-sided [0.48 to 4.02], Standard Error of Mean 0.90

2. Secondary Outcome: Change From Baseline in the CSFQ-14 Total Score at All Other Time Points Assessed
Description: as for outcome 1
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Participants from the FAS, defined as all participants who were randomized and received at least 1 dose of study drug, who had data available for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vortioxetine | Escitalopram
Number analyzed (Participants) | 217 | 207
scores on a scale
  Week 1 (n=213, 206) | 2.5 (0.39) | 2.2 (0.40)
  Week 2 (n=203, 200) | 4.9 (0.46) | 3.7 (0.47)
  Week 4 (n=187, 188) | 7.0 (0.55) | 4.8 (0.55)
  Week 6 (n=175, 176) | 8.0 (0.59) | 6.4 (0.60)

3. Secondary Outcome: Number of Participants With Shifts in the CSFQ-14 From Abnormal to Normal at Each Week Assessed
Description: The CSFQ-14 is a structured self reported questionnaire designed to measure illness- and medication-related changes in sexual functioning consisting of 14 items that measure sexual functioning as a total score (14 items) and on the subscales of pleasure (1 item), desire/frequency (2 items), desire/interest (3 items), arousal (3 items), and orgasm (3 items), rated on an 5 point scale from 1 to 5 with a total score range from 14 to 70. Higher scores reflect higher sexual functioning. Normal sexual functioning is defined as a CSFQ-14 total score of >41 for women and >47 for men. Abnormal sexual functioning is defined as a CSFQ-14 total score of ≤41 for women and ≤47 for men. All subjects entered the study with abnormal sexual functioning. A shift to normal indicates that symptoms have improved.
Time Frame: Baseline and Weeks 1, 2, 4, 6 and 8
Population: Participants from the FAS, defined as all participants who were randomized and received at least 1 dose of study drug, who had data available for this outcome measure. Last observation carried forward.
Measure: Number; unit: number of participants
Arm/Group | Vortioxetine | Escitalopram
Number analyzed (Participants) | 217 | 207
number of participants
  Week 1 (n=213, 205) | 48 | 36
  Week 2 (n=217, 206) | 81 | 63
  Week 4 (n=217, 206) | 93 | 84
  Week 6 (n=217, 206) | 112 | 93
  Week 8 (n=217, 206) | 113 | 91

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug (Up to 12 weeks).
Description: At each visit, the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety analysis set included all participants who received study drug.
Arm/Group | Vortioxetine | Escitalopram
Serious Adverse Events (participants affected / at risk) | 3/224 | 1/221
Other Adverse Events (participants affected / at risk) | 90/224 | 60/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=224) | Escitalopram (N=221)
Angina pectoris (Cardiac disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=224) | Escitalopram (N=221)
Nausea (Gastrointestinal disorders) | 56 | 12
Irritability (General disorders) | 11 | 16
Fatigue (General disorders) | 10 | 12
Headache (Nervous system disorders) | 21 | 17
Dizziness (Nervous system disorders) | 18 | 11
Anxiety (Psychiatric disorders) | 4 | 12
Pruritus generalised (Skin and subcutaneous tissue disorders) | 13 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.